CLINICAL TRIAL: NCT00112684
Title: A Pilot Study of Flavopiridol in Patients With Advanced Solid Tumors
Brief Title: Alvocidib in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00135; NCI-2009-00135 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-2005C0009; CDR0000429582; NCI-7204; OSU-04111; OSU 04111 (Other: Ohio State University Medical Center); 7204 (Other: CTEP); U01CA076576 (NIH); P30CA016058 (NIH); NCT01645540 (obsolete NCT alias)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — alvocidib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, biological therapy) (Experimental): Patients receive alvocidib IV over 4½ hours once weekly in weeks 1-4. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of alvocidib in treating patients with locally advanced or metastatic solid tumors. Drugs used in chemotherapy, such as alvocidib, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Alvocidib may also stimulate the immune system in different ways and stop tumor cells from growing. It may also stop the growth of solid tumors by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxicity profile and dose-limiting toxicity of flavopiridol (alvocidib) in patients with locally advanced or metastatic solid tumors.

II. Determine the maximum tolerated dose of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.

II. Determine the immunomodulatory effects of this drug in these patients. III. Determine pharmacogenomics of this drug, using peripheral blood mononuclear cells, in patients who experience clinical response.

OUTLINE: This is a pilot, dose-escalation study.

Patients receive alvocidib intravenously (IV) over 4½ hours once weekly in weeks 1-4. Treatment repeats every 6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease after 4 courses of therapy discontinue study treatment. Patients who achieve complete remission (CR) receive 1 additional course of therapy beyond documentation of CR. Cohorts of 3-6 patients receive escalating doses of alvocidib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 10 patients are treated at the MTD.

After completion of study treatment, patients are followed within 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor

  * Locally advanced or metastatic disease for which curative treatment does not exist or is no longer effective
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * No previously irradiated* measurable lesion unless lesion demonstrates progressive disease OR there are other measurable lesions outside the irradiated* field
  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
* No uncontrolled brain metastases
* Performance status - ECOG 0-1
* At least 6 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No uncontrolled cardiac arrhythmia
* No uncontrolled hypertension
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to flavopiridol
* No ongoing or active infection
* No uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* More than 12 weeks since prior hepatic arterial chemoembolization
* More than 4 weeks since prior systemic chemotherapy
* No prior flavopiridol
* See Disease Characteristics
* More than 12 weeks since prior radioactive metaiodobenzylguanidine (MIBG)
* More than 4 weeks since prior external beam radiotherapy
* Recovered from all prior tumor-specific therapy
* More than 4 weeks since prior investigational tumor-specific therapy
* Concurrent octreotide for control of carcinoid syndrome allowed
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No other concurrent tumor-specific therapy
* No other concurrent investigational therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-02; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Adverse events of dose escalated alvocidib administered in patients with advanced solid tumors | At weeks 1-4, 7-10, 11 or 12, and within 4 weeks after the completion of study treatment
  Graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.

SECONDARY OUTCOMES:
Pharmacokinetics of alvocidib administered in this schedule | After the first dose of treatment drug
  The pharmacokinetic parameters include Cmax, Css, Clearance, t1/2 α, t1/2 β, central volume of distribution and steady state volume of distribution.
Immunomodulatory effects of alvocidib | Baseline, days 1 and 15 of courses 1 and 2, and within 4 weeks after the completion of study treatment
  Gene expression quantified using Real Time PCR; type 1 and type 2 cytokines, co-stimulatory molecules, and adhesion molecules in PBMCs. Activation of lymphocyte subsets and presence of co-stimulatory and adhesion molecules assessed using multicolor flow cytometry. IL-6 levels in plasma will be measured by ELISA. T-cells will be enriched from PBMCs using mAb-coated immunomagnetic beads and activated with anti-CD3/anti-CD28 mAbs, inomycin or PMA. Cytokine production will be measured using cytometric bead array.
Pharmacogenomics studies on procured PBMCs if clinical responses are observed | Baseline, and within 4 weeks after the completion of study treatment
  Performed if clinical responses are observed. Examine for selected polymorphisms of genes influencing alvocidib metabolism and/or resistance genes that may predict response or toxicity. These changes will be correlated with AUC, toxicity and clinical response to therapy.
Measurement of serum tumor markers depending on the tumor type | Baseline, week 11 or 12, and within 4 weeks after the completion of study treatment
  Markers include CEA, CA 19-9, CA 15-3, PSA, LDH, AFP, b-HCG, pancreastatin, gastrin, pancreatic polypeptide, glucagon, substance-P, neurotensin, calcitonin, somatostatin, vasoactive intestinal peptide, gastrin releasing polypeptide, ACTH, and chromogranin-A.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Shah, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States